CLINICAL TRIAL: NCT04612088
Title: Cognitive Dissonance Based Intervention to Promote Multivitamin Adherence on Bariatric Patients
Brief Title: Intervention for Multivitamin Adherence on Bariatric Patients
Acronym: CDIPMABP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Autonoma de Baja California (Other)
Responsible Party: Principal Investigator, Daniela Lilian Gonzalez Sanchez, Principal Investigator, Universidad Autonoma de Baja California
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D240
Record Dates: First submitted 2020-10-18; First posted 2020-11-02 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Adherence, Medication
Keywords: Adherence; Multivitamin; Bariatric; Gastric Sleeve; Gastric Bypass; Cognitive Dissonance; Intervention
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients will be blindly randomized to one of the two groups and the Cognitive Dissonance doses will be given by two Psychology undergraduate students that are not part of the research team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bariatric Multivitamin (Experimental): Bariatric patients that gave their consent in written will be given a Bariatric Multivitamin containing: Serving Size 2 Tablets: Calories 25, Total Fat 0.5 g, Total Carbohydrates 5g, Total Sugars 2 g, Vitamin A 3,000 mcg, Vitamin C 90 mg, Vitamin D 75 mcg, Vitamin E 100.5 mg, Vitamin K 300 mcg, Thiamin 36 mg, Riboflavin 3.4 mg, Niacin 20 mg, Vitamin B6 4 mg, Folate 1,360 mcg, Vitamin B12 1,000 mcg, Biotin 600 mcg, Pantothenic Acid 20 mg, Calcium 170 mg, Iron 45 mg, Phosphorous 130 mg, Iodine 150 mcg, Magnesium 50 mg, Zinc 16 mg, Selenium 70 mcg, Copper 2 mg, Manganese 2 mg, Chromium 120 mcg, Molybdenum 50 mcg, Sodium 15 mg, Mixed Tocopherols 30 mg, Coenzyme Q10 10 mg and Boron 2 mg.The patients will take 2 tablets once a day for three months.
  Interventions: Behavioral: Cognitive Dissonance
- Waitlist (No Intervention): Bariatric patients that gave their consent in written will be given a Bariatric Multivitamin containing: Serving Size 2 Tablets: Calories 25, Total Fat 0.5 g, Total Carbohydrates 5g, Total Sugars 2 g, Vitamin A 3,000 mcg, Vitamin C 90 mg, Vitamin D 75 mcg, Vitamin E 100.5 mg, Vitamin K 300 mcg, Thiamin 36 mg, Riboflavin 3.4 mg, Niacin 20 mg, Vitamin B6 4 mg, Folate 1,360 mcg, Vitamin B12 1,000 mcg, Biotin 600 mcg, Pantothenic Acid 20 mg, Calcium 170 mg, Iron 45 mg, Phosphorous 130 mg, Iodine 150 mcg, Magnesium 50 mg, Zinc 16 mg, Selenium 70 mcg, Copper 2 mg, Manganese 2 mg, Chromium 120 mcg, Molybdenum 50 mcg, Sodium 15 mg, Mixed Tocopherols 30 mg, Coenzyme Q10 10 mg and Boron 2 mg.The patients will take 2 tablets once a day for three months.

INTERVENTIONS:
Behavioral: Cognitive Dissonance — A blood sample will be taken before the first take of the multivitamins and at the end of the intervention to measure: Hemoglobin, Calcium, Phosphorous, Iron, Copper, Zinc, Vitamin D, and Folate.
  During the three months of the intervention, the intervention group will receive one psycho-educative session and five Cognitive Dissonance sessions.
  Several tests will be applied to the patients at the beginning of the program and after the sessions to measure: patient knowledge and adherence to the multivitamin, self-efficacy, self-care, and Psycho-pathological symptoms.
  The No intervention group on the wait list will receive the five Cognitive Dissonance sessions after the three months of the study.
  Arms: Bariatric Multivitamin

SUMMARY:
This project has a parallel randomized controlled experimental design since within the methodology there will be a control of the conditions under study, that is, the selection of subjects, the way the treatment will be administered, the way in which the observations will be obtained, the use of instruments to perform the measurements and the interpretation of the criteria will be implemented in a homogeneous manner.

Convenience sampling was used to obtain the subjects for the study, the sample size was 34 bariatric patients from a private bariatric center in Tijuana, Baja California, Mexico.

Participants were randomly assigned to one of two groups. The group understudy or experimental or the control group on the waitlist; that is, no researcher or study participant made the decision of treatment that participants receive. The intervention consists of two psychoeducative sessions and five cognitive dissonance sessions. All participants will receive the same multivitamin for the duration of the study. Validated tests for adherence, medication knowledge, self-care, self-efficacy, and psychopathological symptoms were applied to both groups. Additionally, a blood sample was collected for the determination of Hemoglobin, Iron, Copper, Zinc, Calcium, Phosphate, Vitamin D, and Folate. Measurements using tests and blood samples will be made before and after receiving the intervention [pre and post-test]. For results analysis, Repeated measures ANOVA will be used, the study population shall be stratified into subgroups, by type of bariatric surgery, age, and sex; this in order to restrict comparisons to participants who are part of the same subgroup.

The aim of the study is to assess the impact of an intervention based on the cognitive dissonance theory to promote adherence to the bariatric multivitamin.

The hypothesis of the study is: Participants exposed to Festinger's theory-based intervention will exhibit changes in their attitude and behavior towards multivitamin intake as a product of cognitive dissonance.

DETAILED DESCRIPTION:
According to the World Health Organization (WHO), in 2016, 650 million people around the world were already obese, for their part in 2013 the Organization for Economic Cooperation and Development (OCDE) indicated that globally Mexico and the United States had the highest rate of overweight and obesity in adults. Mexico is the second country, after the United States, with the highest obesity, almost one third of Mexican adults (32.4%) suffered from obesity in that year, a significant increase from 24% in 2000.

According to the National Health and Nutrition Survey the states of northern Mexico, as is the case of Baja California, occupy the first places of obesity index nationwide. Morbid Obesity (MO) poses a high health risk in those who suffer from it, as multiple complications arise from it, therefore it is of uttermost importance that this disease is successfully treated and controlled, however, conventional weight loss therapeutics guided by the implementation of behavioral therapy, physical activity, low calorie diet and drug treatment , has shown short-term unsuccessful results. A treatment alternative is Bariatric Surgery (BS) which, according to recommendations issued in 1991 by the U.S. National Institutes of Health (NIH), is considered the treatment of choice for this pathology. While BS has proven to be a successful treatment for long-term sustained weight loss, it is accompanied by major complications such as micronutrient deficiency, which is attributed to intrinsic and extrinsic factors, intrinsic factors refer to deficiencies recorded prior to BS and are related to MO or to the surgical technique itself that induces changes in metabolism in addition to reducing the ability to food in the stomach, limit digestion and cause malabsorption. For their part, extrinsic factors correspond to the lack of adherence in terms of diet and prescribed multivitamin supplementation.

Lack of adherence is related to the level of knowledge about the supplementation and behavior of the morbid patient on decision-making, as they tend to present negative thoughts about the prescribed treatment that are usually accompanied by lack of ability to make changes in both attitude and behavior, which will hardly change even after surgery; this is consistent with the results reported in various studies that indicate that the main behavioral factors of non-adherence to treatment in this population are the low self-efficacy and attitudes that the patient adopts towards treatment on self-care, as well as low self-esteem and distortion of self-concept.

As described, BS can be considered a process of adaptation that can pose a challenge for those who experience it as the person must be aware of the impact of surgery on the body in order to effectively adhere to the agreed treatment plan, making decisions in conjunction with health professionals in order to reduce risk factors , focusing therefore on prevention and timely intervention of them.

In this sense, psychology turns out to be a science that allows to develop instruments that evaluate the congruence between attitudes, thought and behavior, as well as the creation of strategies that promote health promoting the congruence between attitude and behavior. Leon Festinger in 1957 proposed the theory of Cognitive Dissonance, which states that people tend to change their attitudes and behaviors or justify them as a result of the divergence of two cognitions manifested at the same time; according to this theory, the individual strives to achieve consistency within himself. Opinions and attitudes tend to be present in groups that are internally consistent.

Population:

POST-operated Bariatric Surgery patients

Sample:

Post-Bariatric Surgery patients who permanently radiate in the Tijuana Co.

Sampling type:

In the first time, non-probabilistic, convenience sampling for the selection of participants and in a second time for randomization stratification will be performed.

Sampling site:

One private bariatric center in Tijuana, Baja California, Mexico. Research plan

1. Submission and approval of the research protocol to the bioethics committee of the Faculty of Medicine and Psychology (FMYP) of the Autonomous University of Baja California (UABC)
2. Designing the manuals of psycho-educational intervention and dissonance to promote and improve adherence to the multivitamin prescribed in bariatric patients.
3. Once obtaining the bioethics committee approval, the authorities of a private bariatric center operating patients living in Tijuana were consulted to request their cooperation in conducting the research.

(d) Data collection was carried out through the review of clinical records in accordance with the Mexican Official Norm (NOM) NOM-004-SSA3-2012.

(e) Persons who meet the inclusion criteria were contacted by telephone in order to recruit the participants who were included in the study.

(f) Arrange a face-to-face appointment with the person who decides to participate to sign the document "informed consent (IC)" version 1.0, in order to clarify doubts about the methodology of the project and inform him that his participation is voluntary, that at any time he may withdraw his consent and that the information he provides will be handled confidentially, in accordance with NOM-012-SSA3-2012 on Human Research.

(g) Participants were randomly assigned to the experimental group and control group on the waiting list using the on-line tool GraphPad QuickCalcs.

(h) For the application of the measuring instrument (MI) in order to comply with the recommendations of the WHO derived from the COVID pandemic and maintain social distancing, the MI containing all tests was adapted for a digital application using Google Forms and the group sessions were modified to be video conferences through Google Meet.

(i) For the sessions of cognitive dissonance and psycho-education, Psychology Bachelors were trained and randomly assigned to the cognitive or psycho-educational intervention.

(j) The pre-test and post-test blood samples are taken one day after the application of the MI (before and after the intervention), according to NOM-253-SSA1-2012 for the disposal of human blood.

(k) The determination of biomarkers was carried out according to the NOM-007-SSA3-2011 for the operation of clinical laboratories. The analysis of calcium, phosphorus, and serum iron was carried out within the facilities of the UABC Medical Care and Research Centre (CUMAII) using colorimetric spectrophotometry; The levels of Vit-D and Folate were be analyzed by Enzyme-Linked ImmunoSorbent Assay (ELISA), the quantification of hemoglobin was performed during flow cytometry. For the determination of minerals (zinc and copper) in serum, a collaboration agreement will be held with the Graduate Center of the Tijuana Institute of Technology; the method of analysis will be Mass Spectrometry with Inductively Coupled Plasma (ICP/MS).

(l) The week following sampling, 90-minute online intervention sessions will begin every two weeks for three months. It is important to mention that, before the first online session (second week) the participants of both groups will be given a bariatric multivitamin supplement with 60 chewable tablets, dispensing a new one of the same brand as the first, this in order to cover three months of treatment.

(m) Participants were asked to inform through a phone call to the research team in case of presenting any adverse effects such as nausea, vomit, dizziness, or diarrhea. This will be noted in the corresponding document.

(n) Once the post-test data have been obtained, databases will be developed in the SPSS version 26.0 statistical program for Windows, which will be analyzed by repeated-measures ANOVA in order to evaluate the effect of the intervention on adherence to the Multivitamin evidenced by biomarker levels.

ELIGIBILITY:
Inclusion Criteria:

* Nationality: Mexican.
* Place of Residence: City of Tijuana.
* Bariatric techniques: Gastric Sleeve or Bypass Roux in Y.
* Time after surgery: at least 6 months.
* Agree to participate voluntarily by leaving it under signature in the informed consent format.

Exclusion Criteria:

* Nationality: foreign
* Patients who do not reside in the city of Tijuana permanently.
* Bariatric techniques other than Gastric Sleeve or Bypass Roux in Y.
* Time: having passed less than 6 months post-operative.
* Patients who have a cognitive disorder that limits learning or attendance at sessions.
* Patients who are suspended by prescription from vitamin consumption.
* Patients with any post-bariatric surgery complications that are under treatment.
* Patients with a history of alcoholism.
* Pregnant patients.
* Patients who practice high-performance exercise.
* Patients who do not consent to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-04-21 (Estimated); Study Completion 2021-05-24 (Estimated)

PRIMARY OUTCOMES:
Therapy adherence using the MBG (Martin-Bayarre-Grau) Questionnaire | Change from Baseline Adherence level at 3 months
  Adherence of the participants to the multivitamin given, using an instrument validated for the Mexican population. The instrument is based on a Lickert scale, all questions have 5 possible answers that go from Never to Always and have respective values of 0 - 5, the total of the answer points is then recategorized to 0-17 No adherence, 18-37 Partial Adherence, and 38-48 Total Adherence.
Serum Iron, Copper and Zinc levels assessed by Inductively Coupled Plasma Mass Spectroscopy (ICP-MS) | Change from Baseline Iron, Copper and Zinc levels at 3 months
  Participants serum levels of Iron, Copper and Zinc in micrograms per deciliter
Serum Calcium, Phosphate, levels measured by Colorimetric Spectroscopy | Change from Baseline Calcium and Phosphate levels at 3 months
  Participants serum levels of Calcium and Phosphate in milligrams per deciliter
Serum Albumin and Total Protein levels measured by Colorimetric Spectroscopy | Change from Baseline Albumin and Total Protein levels at 3 months
  Participants serum levels of Albumin and Total Protein in grams per deciliter, the Albumin/Globulin Ratio will also be calculated as: Albumin/(Total Protein-Albumin).
Serum Vitamin D and Folate levels measured by Enzyme-Linked ImmunoSorbent Assay (ELISA) | Change from Baseline Vitamin D and Folate levels at 3 months
  Participants serum levels of Vitamin D and Folate in nanograms per mililiter.
Hemoglobin levels measured by the Hematology Analyzer | Change from Baseline Hemoglobin levels at 3 months
  Participants Hemoglobin levels in grams per deciliter will be obtained using an Hematology Analyzer with a Reagent-Less method.

SECONDARY OUTCOMES:
Self-Care Capacity assessed using the Self-care Agency Appreciation (SAA) | Change from Baseline Self-Care levels at 3 months after psychological intervention
  Participants Self-Care Capacity obtained by the Self-care Agency Appreciation (SAA) test that was adapted and validated to be used in Mexican population. The test consists of 24 reagents and aims to assess self-care capabilities by representing all power components.
  The response pattern of this questionnaire includes four options: total disagreement 1, disagreement 2, agreement 3, and total agreement 4. Each individual gets a score ranging from 24 to 112, where the higher the score higher the Self-Care Capacity.
Self-Efficacy assessed using the General Self-Efficacy Scale (GSE) | Change from Baseline Self-Efficacy levels at 3 months after psychological intervention
  Participants level of Self-Efficacy using the validated General Self-Efficacy Scale (GSE), adapted and validated to be used un Mexican population. The test has 10 questions and is based on a Likert scale, with the answer options Not at all true, Hardly true, Moderately true, and Exactly true, each answer scores from 1 to 4. The total score is calculated by finding the sum of the all items. For the GSE, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Psychopathological symptoms assessed using the Symptom Checklist-90-Revised (SCL-90-R) | Change from Baseline Psychopathological symptoms at 3 months after psychological intervention
  Participants referred Psychopathological symptomps will be assessed using the Symptom Checklist-90-Revised (SCL-90-R) which contains the following Symptom Scales: Somatization, Obsessive-Compulsive, Interpersonal Sensitivity, Depression, Anxiety, Hostility, Phobic Anxiety, Paranoid Ideation, Psychoticism and some Global Indices like: Global Severity Index (GSI): Designed to measure overall psychological distress, Positive Symptom Distress Index (PSDI): Designed to measure the intensity of symptoms and Positive Symptom Total (PST): Reports number of self-reported symptoms.
Knowledge of the Multivitaminic supplement assessed using a questionnaire to assess patient knowledge of their medicines | Change from Baseline Knowledge score at 3 months after psychological intervention
  The participants Knowledge of the Multivitaminic supplement will be assessed using a test that consists of 11, open questions that gather the patient's knowledge about the therapeutic objective, the process of use, safety and conservation of the medicines that the patient uses. The answers are evaluated by a pharmacist classifying it as follows Incorrect : Score -1, Does not know: Score 0, Insufficient: Score 1 and Correct: Score 2.
  For the final calculation of total drug knowledge (global PKM) a formula is applied in which each question scored differently based on the conclusions drawn in the different qualitative techniques. The global CPM was categorized into: No knowledge. 0 points, Insufficient knowledge. 0.60 to 1.26 points, Sufficient knowledge. 1.27 to 1.60 points, Optimal knowledge. 1.60 to 2 points.

CONTACTS AND LOCATIONS:
Overall Officials: Gisela Pineda, PhD, Study Director — Professor and Researcher
Locations (1):
- Universidad Autónoma de Baja California, Tijuana, Estado de Baja California, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The data obtained from the Measurement Instrument and Micronutrient levels Pre and Post Intervention as well as all the documents and formats used to make this project will be shared with the research teams that contact us via e-mail.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Study data will be available to be requested for five years after the intervention results have been published on an indexed journal.
Access Criteria: Researchers that wish to obtain our data must contact us via e-mail and provide evidence of their affiliation and research plan.

REFERENCES:
- [Background] Gutiérrez JP, Rivera-Dommarco J, Shamah-Levy T, Villalpando-Hernández S, Franco A, Cuevas-Nasu L, Romero-Martínez M, Hernández-Ávila M. Encuesta Nacional de Salud y Nutrición 2012. Resultados Nacionales. Cuernavaca, México: Instituto Nacional de Salud Pública (MX), 2012.
- [Background] OMS. (2016). WORLD HEALTH STATISTICS MONITORING 2016. In World Health Statistics. https://doi.org/10.1017/CBO9781107415324.004
- [Background] Wimmelmann CL, Dela F, Mortensen EL. Psychological predictors of weight loss after bariatric surgery: a review of the recent research. Obes Res Clin Pract. 2014 Jul-Aug;8(4):e299-313. doi: 10.1016/j.orcp.2013.09.003. Epub 2013 Oct 13. PMID 25091351
- [Background] Gastrointestinal surgery for severe obesity. Consens Statement. 1991 Mar 25-27;9(1):1-20. PMID 1760489
- [Background] Amaya Garcia MJ, Vilchez Lopez FJ, Campos Martin C, Sanchez Vera P, Pereira Cunill JL. [Micronutrients in bariatric surgery]. Nutr Hosp. 2012 Mar-Apr;27(2):349-61. doi: 10.1590/S0212-16112012000200004. Spanish. PMID 22732956
- [Background] Sierra Murguía, M., L, V., & Torres Tamayo, M. (2014). INTERVENCIÓN COGNITIVO-CONDUCTUAL GRUPAL PARA PÉRDIDA DE PESO Y CALIDAD DE VIDA EN PACIENTES CANDIDATOS A CIRUGÍA BARIÁTRICA. Acta Colombiana de Psicología, 17, 25-34.
- [Background] Bergh I, Lundin Kvalem I, Risstad H, Sniehotta FF. Preoperative predictors of adherence to dietary and physical activity recommendations and weight loss one year after surgery. Surg Obes Relat Dis. 2016 May;12(4):910-918. doi: 10.1016/j.soard.2015.11.009. Epub 2015 Dec 1. PMID 26965158
- [Background] Vidal P, Ramon JM, Goday A, Parri A, Crous X, Trillo L, Pera M, Grande L. Lack of adherence to follow-up visits after bariatric surgery: reasons and outcome. Obes Surg. 2014 Feb;24(2):179-83. doi: 10.1007/s11695-013-1094-9. PMID 24101091
- [Background] Sunil S, Santiago VA, Gougeon L, Warwick K, Okrainec A, Hawa R, Sockalingam S. Predictors of Vitamin Adherence After Bariatric Surgery. Obes Surg. 2017 Feb;27(2):416-423. doi: 10.1007/s11695-016-2306-x. PMID 27448232
- [Background] Paredes Despradel, M. E., & Rivero Vergne, A. (2016). Un reto constante: La vida luego de la cirugía bariátrica. Revista Griot, 8(1), 60-72. Recuperado a partir de https://revistas.upr.edu/index.php/griot/article/view/1499
- [Background] Funnell MM, Anderson RM, Ahroni JH. Empowerment and self-management after weight loss surgery. Obes Surg. 2005 Mar;15(3):417-22. doi: 10.1381/0960892053576794. PMID 15826479
- [Background] Festinger, L. (1957). A theory of cognitive dissonance. Stanford University Press.
- [Background] Martín Alfonso, Libertad, & Bayarre Vea, Héctor D., & Grau Ábalo, Jorge A. (2008). Validación del cuestionario MBG (Martín-Bayarre-Grau) para evaluar la adherencia terapéutica en hipertensión arterial. Revista Cubana de Salud Pública, 34(1), .[fecha de Consulta 27 de Octubre de 2020]. ISSN: 0864-3466. Disponible en: https://www.redalyc.org/articulo.oa?id=214/21420865012
- [Background] Weinberg, R. S., Gould, D., & Jackson, A. (1979). Expectations and performance: An empirical test of Bandura's self-efficacy theory. Journal of Sport Psychology, 1(4), 320-331.
- [Background] Rivera Alvarez LN. [Self-care agency ability in people suffering from high blood pressure hospitalised in Bogota, Colombia]. Rev Salud Publica (Bogota). 2006 Sep-Dec;8(3):235-47. doi: 10.1590/s0124-00642006000300009. Spanish. PMID 17269223
- [Background] Garcia Delgado P, Gastelurrutia Garralda MA, Baena Parejo MI, Fisac Lozano F, Martinez Martinez F. [Validation of a questionnaire to assess patient knowledge of their medicines]. Aten Primaria. 2009 Dec;41(12):661-8. doi: 10.1016/j.aprim.2009.03.011. Epub 2009 May 29. Spanish. PMID 19481298
- [Background] Banik A, Schwarzer R, Knoll N, Czekierda K, Luszczynska A. Self-efficacy and quality of life among people with cardiovascular diseases: A meta-analysis. Rehabil Psychol. 2018 May;63(2):295-312. doi: 10.1037/rep0000199. PMID 29878834
- [Background] Modi AC, Zeller MH, Xanthakos SA, Jenkins TM, Inge TH. Adherence to vitamin supplementation following adolescent bariatric surgery. Obesity (Silver Spring). 2013 Mar;21(3):E190-5. doi: 10.1002/oby.20031. PMID 23404956
- [Background] Parrott J, Frank L, Rabena R, Craggs-Dino L, Isom KA, Greiman L. American Society for Metabolic and Bariatric Surgery Integrated Health Nutritional Guidelines for the Surgical Weight Loss Patient 2016 Update: Micronutrients. Surg Obes Relat Dis. 2017 May;13(5):727-741. doi: 10.1016/j.soard.2016.12.018. Epub 2017 Jan 19. PMID 28392254
- [Background] Savino, P., Carvajal, C., Nassar, R., & Zundel, N. (2013). Necesidades nutricionales específicas después de cirugía bariátrica: Specific nutritional requirements following bariatric surgery. Revista Colombiana de Cirugía, 28(2), 161-171. http://www.scielo.org.co/scielo.php?script=sci_arttext&pid=S2011-75822013000200009&lng=en&nrm=iso&tlng=
- [Background] Kalarchian MA, Marcus MD. Psychosocial Interventions Pre and Post Bariatric Surgery. Eur Eat Disord Rev. 2015 Nov;23(6):457-62. doi: 10.1002/erv.2392. Epub 2015 Sep 14. PMID 26364715
- [Background] Mahawar KK, Clare K, O'Kane M, Graham Y, Callejas-Diaz L, Carr WRJ. Patient Perspectives on Adherence with Micronutrient Supplementation After Bariatric Surgery. Obes Surg. 2019 May;29(5):1551-1556. doi: 10.1007/s11695-019-03711-z. PMID 30652245
- [Background] Derogatis LR, Lipman RS, Covi L. SCL-90: an outpatient psychiatric rating scale--preliminary report. Psychopharmacol Bull. 1973 Jan;9(1):13-28. No abstract available. PMID 4682398